CLINICAL TRIAL: NCT00646685
Title: Prospective Randomized Trial for Comparison of Duct-to-duct and Roux-en-y Hepaticojejunostomy for Biliary Reconstruction in Adult Living Donor Liver Transplantation
Brief Title: Duct-to-duct vs Roux-en-y Hepaticojejunostomy for Biliary Reconstruction in Adult Living Donor Liver Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-0498-B
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2012-06

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other)
  Interventions: Procedure: surgical technique: duct-to-duct biliary reconstruction
- 2 (Other)
  Interventions: Procedure: surgical technique: roux-en-y biliary reconstruction

INTERVENTIONS:
Procedure: surgical technique: duct-to-duct biliary reconstruction — surgical reconstruction
  Arms: 1
Procedure: surgical technique: roux-en-y biliary reconstruction — surgical reconstruction
  Arms: 2

SUMMARY:
The purpose of this study is to empirically determine whether one of 2 surgical techniques commonly used for bile duct reconstruction during living donor liver transplantation results in fewer biliary complications. Also, this study may identify patient group(s) that particularly benefit from a particular technique.

DETAILED DESCRIPTION:
The purpose of this study is to compare the incidence of biliary complications (bile leaks and strictures) following duct-to-duct and roux-en-y biliary reconstruction during right lobe living donor liver transplantation.

Biliary complications are much more common with right lobe living donor liver grafts than with whole organ grafts and are considered a major limitation of this surgery. Two surgical techniques are currently used for biliary reconstruction and each has its advantages/disadvantages. However, it is unclear which technique leads to fewer biliary complications. Retrospective studies which examine biliary complication rates may be hampered by such factors as a surgeon's bias or inexperience with a particular technique. Therefore a prospective randomized trial is needed.

ELIGIBILITY:
Inclusion Criteria:

* patient with end-stage liver disease
* living donor liver transplantation using right hemi-liver as graft
* duct anastomosis possible at time of surgery
* donor and recipient aged 18 yrs or older
* written informed consent obtained

Exclusion Criteria:

* duct anastomosis not possible
* acute fulminant liver failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-02; Primary Completion 2015-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Biliary complications defined as leaks and strictures within the first year post LDLT; | 1 year

SECONDARY OUTCOMES:
Graft and patient survival | 1 year post-transplant
Length of hospital-stay and ICU-stay | within first 30 days after discharge
Any infection or rejection episodes | 1 year post- transplant
time to full oral nutrition | within 30 days of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Markus Selzner, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada